CLINICAL TRIAL: NCT03416556
Title: The Initial Effects on Pain, Pain Sensitivity, Range of Motion and Muscle Strength of an Anteroposterior Mobilization of the Glenohumeral Joint in Overhead Athletes With Chronic Shoulder Pain
Brief Title: Manual Therapy in Chronic Shoulder Pain Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Professor, University of Alcala
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H1496053548524
Record Dates: First submitted 2018-01-11; First posted 2018-01-31 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: * The participant were assigned to the treatment group with a computer program.
  * Outcomes assessor did´t know the treatment applied to the participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mobilization to the glenohumeral joint (Experimental): This condition consisted on the application of a passive rhythmic AP mobilization to the glenohumeral joint of the affected shoulder
  Interventions: Procedure: Mobilization to the glenohumeral joint
- The manual contact condition (Sham Comparator): In this condition the therapist positioned the patient in a mid-range position of glenohumeral abduction and internal rotation and applied the hands to the same contact point as in the treatment condition.
  Interventions: Procedure: The manual contact condition; Other: No-contact condition
- No-contact condition (No Intervention): There was no manual contact between the therapist and the participant

INTERVENTIONS:
Procedure: Mobilization to the glenohumeral joint — The treatment condition consisted on the application of a passive rhythmic AP mobilization to the glenohumeral joint of the affected shoulder. In particular, a Grade III AP glide to the humeral head with the arm positioned in 90º of glenohumeral abduction and full internal rotation was used. The posterior gliding force to the humeral head was applied maintaining the glide at right angles to the plane of movement and at a frequency of 2 Hz which was controlled by means of a metronome. The arm was returned to its original position between each set.
  Other Names: Joint Manipulation
  Arms: Mobilization to the glenohumeral joint
Procedure: The manual contact condition — During the manual contact condition the therapist positioned the patient in a mid-range position of glenohumeral abduction and internal rotation and applied the hands to the same contact point as in the treatment condition. However, a simulated posterior glide was performed but with minimal pressure actually applied. The number of repetitions and sets were as per the treatment condition.
  Arms: The manual contact condition
Other: No-contact condition — During the no-contact condition, the subject remained in the initial starting position thorough the entire session but there was no manual contact between the therapist and the participant. The total treatment time was the same as per the other conditions.
  Arms: The manual contact condition

SUMMARY:
Background: Passive oscillatory mobilizations are often employed by physiotherapists to reduce shoulder pain and increase function. However, there is little data about the neurophysiological effects of these mobilizations.

Objectives: To investigate the initial effects of an anteroposterior (AP) shoulder joint mobilization on measures of pain and function in overhead athletes with chronic shoulder pain.

DETAILED DESCRIPTION:
Design: Double-blind, controlled, within-subjects repeated-measures design Method: Thirty-one overhead athletes with chronic shoulder pain participated. The effects of a 9-min, AP mobilization of the glenohumeral joint were compared with manual contact and no-contact interventions. Pressure pain threshold (PPT), range of movement (ROM), muscle strength, self-reported pain, and disability were measured immediately before and after each intervention.

ELIGIBILITY:
Inclusion Criteria:

* History of chronic shoulder pain lasting ≥3 months.
* Play overhead sport regularly.

Exclusion Criteria:

* Had a non-musculoskeletal origin of shoulder pain.
* Previous surgery to the shoulder complex.
* Frozen shoulder.
* Any co-existing inflammatory, infectious or neurological condition.
* The patient from physiotherapy treatment.
* Any evidence of pain referred from the cervical spine to the shoulder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Self-reported shoulder pain | Change from Baseline at 5 minutes after intervention
  Participants were asked to indicate the intensity of their current shoulder pain using a numeric rating pain scale (NRPS). In this scale, 0 is not pain and 10 is the worse pain possible

SECONDARY OUTCOMES:
Shoulder disability | Change from Baseline at 24 hours after treatment
  The DASH is comprised of 30 items (disability/symptom section) and two optional sections related to the impact of pathology on work and sports. Each item is scored from 1 to 5 with increasing values representing more severity of symptoms. The total score for the disability/symptoms section ranges from 30 to 150, but it is then transformed to a scale from 0 (better score possible) to 100 (worse score possible).
Shoulder range of movement (ROM) | Change from Baseline at and 5 minutes after treatment
  Active elevation in the scapular plane and passive glenohumeral internal and external rotation were measured using a Standard BASELINE ® 12-inch plastic goniometer following previous guidelines. The 0 degrees of movement is worse and 180 degrees is the better
Shoulder muscles strength | Change from Baseline at 5 minutes after treatment
  Isometric strength of the shoulder internal and external rotator musculature was measured using a portable hand-held dynamometer (Nicholas Manual Muscle Tester, Lafayette Instruments, USA). Normal external rotation strength is 20 Newtons and 27 newton in internal rotation strength
Pressure pain threshold (PPT) | Change from Baseline at 5 minutes after treatment
  The PPT was measured using an analogue Fisher algometer (Force Dial model FDK, Wagner Instruments) with a surface area at the round tip of 1cm2. The algometer probe tip was applied perpendicular to the skin at a rate of 1kg/cm2/s until the first onset of pain. The PPT value is specific in each subject.The minimal clinically important difference is 2Kg/cm

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pecos-Martin, Dr, Principal Investigator — Alcala University
Locations (1):
- Clinical University, Alcalá de Henares, Madrid, Spain

DOCUMENTS (1):
  • Study Protocol (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT03416556/Prot_000.pdf